CLINICAL TRIAL: NCT00613015
Title: Interdisciplinary Medication Development for Multiple Risk Factors in Relapse.
Brief Title: Stress and Medication Effects on Cocaine Cue Reactivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R01DA021690 (NIH); R01DA021690 (NIH)
Record Dates: First submitted 2008-02-08; First posted 2008-02-12 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Cocaine Related Disorders
Keywords: Cocaine Addiction; Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Guanfacine; Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Modafinil/Stress (Experimental): Participants received placebo for 2 days. modafinil on the third day and participated in the TRIER social stress task on the third day.
  Interventions: Drug: Modafinil
- Modafinil/no stress (Experimental): Participants received placebo for 2 days. modafinil on the third day and did not participate in the TRIER social stress task on the third day.
  Interventions: Drug: Modafinil
- Guanfacine/stress (Experimental): Participants received guanfacine for 3 days and participated in the TRIER social stress task on the third day.
  Interventions: Drug: Guanfacine
- Guanfacine/no stress (Experimental): Participants received guanfacine for 3 days and did not participate in the TRIER social stress task on the third day.
  Interventions: Drug: Guanfacine
- Placebo/Stress (Placebo Comparator): Participants received placebo for 3 days and participated in the TRIER social stress task on the third day.
  Interventions: Drug: Placebo
- Placebo/no stress (Placebo Comparator): Participants received placebo for 3 days and did not participate in the TRIER social stress task on the third day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine
  Arms: Guanfacine/no stress; Guanfacine/stress
Drug: Modafinil
  Arms: Modafinil/Stress; Modafinil/no stress
Drug: Placebo
  Arms: Placebo/Stress; Placebo/no stress

SUMMARY:
Stressful situations and cues associated with cocaine can lead to craving in cocaine dependent individuals. The purpose of this study is to determine whether guanfacine or modafinil are effective in reducing stress and cue induced craving in cocaine dependent individuals.

DETAILED DESCRIPTION:
Stress and cocaine cues produce craving and ultimately relapse in cocaine dependent individuals. This is a randomized, double-blind, placebo-controlled study evaluating the effects of either guanfacine (Tenex) or modafinil (Provigil) on stress and cue induced craving in cocaine dependent individuals. Cocaine dependence will be assessed in adults (ages 18-65) as defined by DSM-IV criteria. If the subject signs the consent form, meets the study criteria and does not meet the exclusion criteria they will be included in the study. Subjects will report to the General Clinical Research Center (GCRC) at the Medical University of South Carolina (MUSC), for an outpatient visit and will receive their first dose of study medication. The following day subjects will return to the GCRC and admitted for the duration of the study (two days and one night). There will be a one-week and a one-month follow-up visit. Subjects will be randomly assigned to one of two treatment groups (guanfacine or placebo). Each subject will also be randomly assigned to either a stress or no-stress subgroup. On the test day (day 3) subjects in the stress group will be asked to perform a speech and a math problem in front of an audience (Trier Social Stress Test, TSST), while the no-stress group will be asked to sit quietly and read. Following these tasks, each subject will be exposed to neutral (control) cues and immediately afterwards the subjects will be exposed to cocaine cues (cocaine paraphernalia). Craving/mood, physiological activity, and endocrine responses, will be assessed at pre-set intervals throughout the testing procedure. The cue reactivity protocol will be repeated on the one-week follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.

Subjects must consent to remain abstinent from all drugs of abuse (except nicotine) during the GCRC admission.

Because of the high comorbidity of alcohol and marijuana use and cocaine dependence, individuals meeting dependence for alcohol and marijuana will be included. Individuals requiring medical detox from alcohol will be excluded.

Subjects must consent to random assignment to stress vs. no stress and drug treatment conditions.

Exclusion Criteria:

Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control. Modafinil inhibits metabolism of steroidal contraceptives via CYP3A4 and can reduce the effectiveness of this type of birth control, female subjects must use one of the following methods of birth control: barrier methods (diaphragm or condoms with spermicide or both), surgical sterilization, use of an intra-uterine contraceptive device, or complete abstinence from sexual intercourse.

Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular (including but not limited to left ventricular hypertrophy (unless a cardiologist deems that it is not clinically significant), mitral valve prolapse, left bundle branch block, myocardial infarction, and angina), pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect HPA axis function.

Subjects with any liver function test (LFTs) of greater than two times normal, as compromised liver function can interfere with HPA axis activity (Williams and Dluhy 1987) and may affect drug metabolism.

Subjects with Addison's disease, Cushing's disease or other diseases of the adrenal cortex likely to affect HPA axis function.

Subjects with a history of or current psychotic disorder or bipolar affective disorder as these may interfere with HPA function.

Subjects with current major depressive disorder or post-traumatic stress disorder as these disorders are associated with characteristic changes in HPA axis function.

Subjects receiving synthetic glucocorticoid therapy, any exogenous steroid therapy, or treatment with other agents that interfere with HPA axis function within one month of the time of testing.

Subjects taking any psychotropic medications, opiates or opiate antagonists because these may affect HPA axis function.Participants taking SSRI's will be included.

Subjects required to take medications that could adversely interact with study medications, including, but not limited to, azole type antifungals, cyclosporine, warfarin, theophylline, or carbamazepine. Any medications that induce or inhibit CYP3A4 pathways are excluded, as modafinil is metabolized through this enzyme system.

Subjects with any acute illness or fever as this may affect HPA axis activity. Individuals who otherwise meet study criteria will be rescheduled for evaluation for participation.

Subjects who are grossly obese (BMI > 39), as this may interfere with HPA axis function.

Subjects who are unwilling or unable to maintain abstinence from alcohol and other drugs of abuse (except nicotine) prior to the stress task procedure.

Subjects meeting DSM-IV criteria for substance dependence (other than nicotine, cocaine, alcohol or marijuana) within the past 60 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2008-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E See, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina-GCRC, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between April 2008 and May 2012. Participants were primarily recruited through newspaper and television advertisements and respondent driven sampling. All study procedures took place at the Medical University of South Carolina.
Pre-assignment Details: 50 participants were enrolled and dropped for unknown reason. 22 participants were enrolled but failed the urine drug screen. 2 participants were unable to complete due to obtaining employment. 2 participants completed procedures, but were later discovered to have bipolar disorder. Their data was not used.
Groups:
- Modafinil/Stress: Participants received Modafinil for three days and completed a TRIER social stress task on the third day.
- Modafinil/No Stress: Participants received modafinil for 3 days and did not complete the TRIER social stress task on the third day.
- Guanfacine/Stress: Participants received placebo for 2 days, guanfacine for 1 day, and completed the TRIER social stress task on the third day.
- Guanfacine/No Stress: Participants received placebo for 2 days, guanfacine for 1 day, and did not complete the TRIER social stress task on the third day.
- Placebo/Stress: Participants received placebo for 3 days and completed the TRIER social stress task on the third day.
- Placebo/No Stress: Participants received placebo for 3 days and did not complete the TRIER social stress task on the third day.
Period: Overall Study
Arm/Group | Modafinil/Stress | Modafinil/No Stress | Guanfacine/Stress | Guanfacine/No Stress | Placebo/Stress | Placebo/No Stress
Started | 13 | 12 | 26 | 24 | 15 | 19
Completed | 13 | 11 (One participant did not complete the one-week follow-up visit.) | 23 (Three participants did not complete one-week follow-up visit.) | 21 (Three participants did not complete one-week follow-up visit.) | 13 (Two participants did not complete one-week follow-up visit.) | 16 (Three participants did not complete one-week follow-up visit.)
Not Completed | 0 | 1 | 3 | 3 | 2 | 3
Not completed — Lost to Follow-up | 0 | 1 | 3 | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil/Stress | Modafinil/No Stress | Guanfacine/Stress | Guanfacine/No Stress | Placebo/Stress | Placebo/No Stress | Total
Number analyzed (Participants) | 13 | 12 | 26 | 24 | 15 | 19 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 26 | 24 | 15 | 19 | 109
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.46 (8.03) | 38.5 (10.49) | 41 (10.05) | 40.92 (9.55) | 40.2 (9.13) | 44 (8.6) | 41.41 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 4 | 3 | 5 | 19
  Male | 10 | 9 | 25 | 20 | 12 | 14 | 90
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 26 | 24 | 15 | 19 | 109

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Craving
Description: Participants were randomized to the modafinil, guanfacine, or placebo treatment group. Participants were then randomized to participate in the TRIER social stress task or to read magazines for 15 minutes. Following the task, participants were exposed to neutral cues for 2 minutes and cocaine cues for 2 minutes. Immediately following the cocaine cue exposure, participants were asked to rate cocaine craving on a 10-point Likert scale, with 0 being Not at All and 10 being Extremely.
Time Frame: Post Trier social stress task + Cocaine Cue 2:30 pm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modafinil/Stress | Modafinil/No Stress | Guanfacine/Stress | Guanfacine/No Stress | Placebo/Stress | Placebo/No Stress
Number analyzed (Participants) | 13 | 12 | 26 | 24 | 15 | 19
units on a scale | 3.08 (3.59) | 4.36 (2.84) | 1.54 (3.06) | 3.13 (3.49) | 1.8 (2.8) | 2.11 (2.4)

2. Secondary Outcome: Cortisol- 2:30 pm, Immediately Following Trier Social Stress Task + Cocaine Cue Exposure
Description: Participants were randomized to receive to the modafinil, guanfacine, or placebo treatment group. Participants were then randomized to complete a TRIER social stress task or read magazines for 15 minutes. Following the task, participants were exposed to neutral cues for two minutes and control cues for two minutes. Immediately following exposure to the cocaine cue, saliva samples were collected to measure cortisol levels.
Time Frame: Immediately following trier + cocaine cue exposure
Measure: Mean (Standard Deviation); unit: mcg/dl
Arm/Group | Modafinil/Stress | Modafinil/No Stress | Guanfacine/Stress | Guanfacine/No Stress | Placebo/Stress | Placebo/No Stress
Number analyzed (Participants) | 13 | 12 | 26 | 24 | 15 | 19
mcg/dl | 12.55 (3.27) | 11.69 (5.57) | 13.19 (5.36) | 9.06 (2.19) | 12.42 (3.95) | 8.94 (2.48)

ADVERSE EVENTS:
Arm/Group | Modafinil/Stress | Modafinil/No Stress | Guanfacine/Stress | Guanfacine/No Stress | Placebo/Stress | Placebo/No Stress
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/26 | 0/24 | 0/15 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/26 | 0/24 | 0/15 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No